CLINICAL TRIAL: NCT03967470
Title: Bacteriotherapy to Improve Underarm Odor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CMET
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Bromhidrosis
MeSH Terms: conditions — Body Odor

STUDY DESIGN:
Intervention Model Description: two groups of 30 people, one month of bacterial spray use and the other month placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Double blind: participants nor outcome assessors, odor panel or care providers do not know which spray they use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo arm (Placebo Comparator): Placebo spray used during one month
  Interventions: Biological: Bacterial spray
- Treatment arm (Active Comparator): Bacteria spray used during one month
  Interventions: Biological: Bacterial spray

INTERVENTIONS:
Biological: Bacterial spray — Bacterial spray containing bacteria that do not cause underarm malodor

SUMMARY:
The goal is to improve the underarm odor by changing the microbiome. The autochthonous bacterial community is replaced by a non-smelling microbiome, by daily application of bacteria in a spray.

DETAILED DESCRIPTION:
Participants are recruited and selected based on their initial underarm odor and underarm microbiome. The participants use two sprays: one spray containing the bacteria, and the other nothing (placebo). Participants do not know which spray they have. They use one spray during one month, and meanwhile take samples of their underarm microbiome (for sequencing), volatome (for GC/MS analysis) and odor (for odor panel analysis). Samples are stored in the freezer and brought to the university after one month, when they receive the second spray. The bacterial spray contains bacteria that are correlated with good underarm odor.

ELIGIBILITY:
Inclusion Criteria:

* above average underarm malodor
* microbiome dominated with malodorous bacteria

Exclusion Criteria:

* not healthy
* microbiome with too high levels of Staphylococcus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Improved underarm odor | 1 month
  Odor panel and GC/MS results provide insights on underarm odor development

CONTACTS AND LOCATIONS:
Overall Officials: Tom Van de Wiele, PhD, Study Chair — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
All data remain confidential

REFERENCES:
- [Result] Callewaert C, Lambert J, Van de Wiele T. Towards a bacterial treatment for armpit malodour. Exp Dermatol. 2017 May;26(5):388-391. doi: 10.1111/exd.13259. Epub 2017 Feb 2. PMID 27892611
- See also: Related Info — http://www.drarmpit.com